CLINICAL TRIAL: NCT05179460
Title: Post-authorization Safety Study and Real-world Evaluation of the Use of Pentosan Polysulfate Sodium and the Development of Pigmentary Maculopathy and Pigmentary Retinopathy
Brief Title: A Study of Pentosan Polysulfate Sodium and the Development of Pigmentary Maculopathy and Pigmentary Retinopathy
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109142; RWJ800077ICS4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-12-10; First posted 2022-01-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pigmentary Maculopathy; Pigmentary Retinopathy; Interstitial Cystitis
MeSH Terms: conditions — Retinitis Pigmentosa; Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clean Cohort: Clean cohort refers to cohort of participants who had their first documented exposure to pentosan polysulfate sodium (PPS; Elmiron) on or after 22 May 2018 and who are assumed to have had shorter exposure (the earliest available data based on the linked database between the IRIS registry and Komodo database in this study).
- Overall Cohort: Overall cohort refers to cohort of participants who had their first documented exposure to PPS (Elmiron) any time beginning 01 January 2015 and who are assumed to have relatively longer exposure (the earliest available data based on the linked database between the intelligent research in sight (IRIS) registry and Komodo database in this study).
- Interstitial Cystitis (IC) Cohort: IC cohort refers to cohort of participants who had at least one IC diagnosis beginning 01 January 2015 and had no documented exposure to PPS based on the records from the Komodo database (the earliest available data based on the linked database between the IRIS registry and Komodo database in this study).

SUMMARY:
The purpose of this study is to evaluate incidence and prevalence rates of the study endpoints (pigmentary maculopathy [PM]/ pigmentary retinopathy [PR]/Any, PM/PR/ pentosan polysulfate sodium [PPS], and PM/PR/Non-PPS) in relation to PPS exposure, and in participants with interstitial cystitis (IC) but not exposed to PPS; changes in visual acuity (VA) over time; participant treatment journey leading to PPS treatment, and potential risk factors associated with the occurrence of PM/PR/PPS.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at least 6 months baseline information prior to index date (this may apply to the relevant databases, if the study participants are identified and the outcomes are ascertained via multiple linked data source) For the pentosan polysulfate sodium (PPS) Cohort
* Participants must have records in both the intelligent research in sight (IRIS) database and the closed claims portion of the Komodo claims database and have at least one record of PPS dispensing For the interstitial cystitis (IC) Cohort not exposed to PPS
* Participants must have records in both the IRIS database and the closed claims portion of the claims database; have at least one diagnosis of IC; and have no record of PPS dispensing

Exclusion Criteria:

- Evaluated based on the Komodo database. Participants will be excluded from the study if they have no information on age or sex (or both)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is derived from the United States-based electronic databases, including the Intelligent Research in Sight (IRIS) Registry, American Urological Association Quality (AQUA) Registry, and Komodo Health claims. The selection of the study participants and cohort creation will be determined by the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Clean Cohort: Incidence Rate of Pigmentary Maculopathy (PM)/ Pigmentary Retinopathy (PR)/Any Cases | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants exposed to pentosan polysulfate sodium [PPS]). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases divided by number of person-years time at risk.
Clean Cohort: Incidence Rate of PM/PR/PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants exposed to PPS). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases divided by number of person-years time at risk.
Clean Cohort: Incidence Rate of PM/PR/Non-PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants not exposed to PPS). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases divided by number of person-years time at risk.
Clean Cohort: Prevalence Rate of PM/PR/Any Cases | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Prevalence rate is defined as number of prevalent cases per number of target cohort assessed (example, number of participants exposed to PPS).
Clean Cohort: Prevalence Rate of PM/PR/PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Prevalence rate is defined as number of prevalent cases per number of target cohort assessed (example, number of participants exposed to PPS).
Clean Cohort: Prevalence Rate of PM/PR/Non-PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Prevalence rate is defined as number of prevalent cases per number of target cohort assessed (example, number of participants not exposed to PPS).
Overall Cohort: Incidence Rate of PM/PR/Any Cases | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants exposed to pentosan polysulfate sodium [PPS]). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases divided by number of person-years time at risk.
Overall Cohort: Prevalence Rate of PM/PR/Any Cases | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Prevalence rate is defined as number of prevalent cases per number of target cohort assessed (example, number of participants exposed to PPS).
Overall Cohort: Incidence Rate of PM/PR/PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants exposed to pentosan polysulfate sodium [PPS]). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases divided by number of person-years time at risk.
Overall Cohort: Prevalence Rate of PM/PR/PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Prevalence rate is defined as number of prevalent cases per number of target cohort assessed (example, number of participants exposed to PPS).
Overall Cohort: Number of PM/PR/PPS Cases Among the PM/PR/Any Cases | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Number of PM/PR/PPS cases among the PM/PR/any cases will be reported.
Clean Cohort: Change in Visual Acuity (VA) in Relation to PPS Dose | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Change in VA in relation to PPS dose will be reported. It will be assessed based on the following categories: a) No change (refers to less than [<] 1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) greater than or equal to (>=) 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Clean Cohort: Change in VA in Relation to PM/PR/Any Cases | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/Any) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Clean Cohort: Change in VA in Relation to PM/PR/PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/PPS) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Clean Cohorts: Change in VA in Relation to PM/PR/Non-PPS | Data analysed retrospectively from 22-May-2018 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/Non-PPS) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Overall Cohort: Change in Visual Acuity (VA) in Relation to PPS Dose | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA in relation to PPS dose will be reported. It will be assessed based on the following categories: a) No change (refers to less than [<] 1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) greater than or equal to (>=) 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Overall Cohort: Change in VA in Relation to PM/PR/Any Cases | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/Any) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Overall Cohort: Change in VA in Relation to PM/PR/PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/PPS) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Overall Cohort: Change in VA in Relation to PM/PR/Non-PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/Non-PPS) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
Interstitial Cystitis (IC) Cohort: Incidence Rate of PM/PR/Any Cases Among the Participants with IC and No-Exposure to PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Incidence rate is defined as number of incident cases per number of all participants at risk (that is, number of all participants not exposed to PPS). Incidence rate is calculated by using formula: incidence rate (per 100 person-years)= number of incidence cases per number of person-years time at risk.
IC Cohort: Change in VA in Relation to PM/PR/Any Cases | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA in relation to study endpoint (PM/PR/Any) will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
IC Cohort: Change in VA Based on Age | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA based on age among participants exposed to PPS and without exposure to PPS will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
IC Cohort: Change in VA Based on Sex | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA based on sex among participants exposed to PPS and without exposure to PPS will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.
IC Cohort: Change in VA Based on Time Between the First and Last VA Measurement in Matched Cohorts | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Change in VA based on time between the first and last VA measurement in matched cohorts among participants exposed to PPS and without exposure to PPS will be reported. It will be assessed based on the following categories: a) No change (refers to <1 line of worsening or improvement, considered not clinically meaningful); b) 1 to <3 lines of worsening; c) >= 3 lines of worsening; d) 1 to <3 lines of improvement; e) >= 3 lines of improvement.

SECONDARY OUTCOMES:
Demographic characteristics of Cohorts: Age | Baseline
  Demographic characteristics of cohorts (age) will be reported.
Demographic characteristics of Cohorts: Sex | Baseline
  Demographic characteristics of cohorts (sex) will be reported.
Demographic characteristics of Cohorts: Race | Baseline
  Demographic characteristics of cohorts (race including Asian, black or African American, other, White or Caucasian) will be reported.
Demographic characteristics of Cohorts: Ethnicity | Baseline
  Demographic characteristics of cohorts (ethnicity including Hispanic and non-Hispanic) will be reported.
Number of Participants with Comorbidities | Baseline
  Number of participants with general comorbidities (diabetes, hypertension, hypercholesterolemia, vaginitis, urinary tract infection [UTI], detrusor instability, urge incontinence, and overactive bladder, autoimmune disease, Malignant tumor(s) of head and neck [plus documentation of radiation therapy] and Radiation cystitis) and ocular comorbidities (diabetic retinopathy, diabetic macular edema, optic neuropathy, glaucoma, glaucoma-related procedure, cataract [diagnosis], cataract [procedure]) will be reported.
Number of Participants who had Provider Characteristics | Baseline
  Number of participants who had provider characteristics (treating provider specialty [retina specialist, non-retina specialist, general ophthalmologist, optometrist]; rural or non-rural location of index practice [rural/non-rural; United States Department of Agriculture Economic research service 2010 classification]) will be reported.
Overall Cohort: Distribution of International Classification of Diseases (ICD)-9/10 Codes | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  ICD-9/10 codes are compared among the participants who are exposed to PPS will be reported.
Participant's Journey to PPS | Data analysed retrospectively from 01-Jan-2015 to 31-Mar-2021 will be examined
  Participant's journey to PPS is defined as the sequence of medications and other interventions the participant received before and after receiving PPS.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen R&D, LLC, Titusville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted CSR synopsis-RWJ800077ICS4001 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR109142&attachmentIdentifier=ac80f1d9-8a10-42fa-bf31-34ddaf831f62&fileName=REDACTED_CSR-Synopsis-RWJ800077ICS4001-1180982.pdf&versionIdentifier=